CLINICAL TRIAL: NCT03223792
Title: Acceptance Of A Partially-Hydrolyzed Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3389-1
Record Dates: First submitted 2017-07-12; First posted 2017-07-21 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Stool

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Other: Control
- Investigational (Experimental)
  Interventions: Other: Investigational

INTERVENTIONS:
Other: Control — Routine cow's milk-based infant formula
  Arms: Control
Other: Investigational — Partially-hydrolyzed cow's milk protein infant formula
  Arms: Investigational

SUMMARY:
This clinical trial will evaluate stool consistency in infants receiving one of two study formulas through a 14-day feeding period.

ELIGIBILITY:
Inclusion Criteria:

* Singleton 28-300 days of age at randomization
* Gestational age less than or equal to 35 weeks
* Receiving minimum 18oz infant formula in the 24hrs prior to randomization
* History of hard stools or stooling difficulty
* Signed informed consent and protected health information

Exclusion Criteria:

* Current diagnosis of cow's milk protein allergy or intolerance
* Use of extensively hydrolyzed or amino acid formula at randomization
* Any abdominal or gastrointestinal surgery prior to randomization
* History of underlying metabolic or chronic disease or congenital malformation
* Organic causes of constipation

Ages: 28 Days to 300 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Stool consistency measured by MJN stool consistency scale | 14 days

SECONDARY OUTCOMES:
Stool frequency | 14 days
Formula acceptance measured by intake diary | 14 days
Formula gastrointestinal tolerance measured by diary | 14 days
Bowel movement characteristics by diary | 14 days
Medically confirmed adverse events throughout the study period | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Wu, Study Director — Mead Johnson Nutrition
Locations (11):
- United States (11):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Deaconess Clinical Research, Evansville, Indiana
  - Deaconess Clinic, Newburgh, Indiana
  - Kentucky Pediatrics/Adult Research, Bardstown, Kentucky
  - Owensboro Pediatrics, Owensboro, Kentucky
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Coastal Pediatric Research, Charleston, South Carolina
  - DCOL Center for Clinical Research, Longview, Texas

IPD SHARING:
Plan to Share IPD: No